CLINICAL TRIAL: NCT04868474
Title: Combining Default Choices and a Decision Aid to Improve Tobacco Cessation at 6 Months in Primary Care Patients: a Pragmatic, Cluster-randomized Trial
Brief Title: Combining Default Choices and a Decision Aid to Improve Tobacco Cessation
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: Tobacco Control Fund Switzerland (Other Government); Swiss Medical Association (FMH) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FIRST
Record Dates: First submitted 2021-03-03; First posted 2021-05-03 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation
Keywords: Behavioral economics; Shared decision making; Default choice; Primary care
MeSH Terms: conditions — Smoking Cessation | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Who Masked: Participant
Masking Description: The smoking cessation experts administering the trainings will not be blinded. GPs will be not be blinded. GPs in the control group will likely realize their training is shorter, and GPs in the intervention group will realize their training is different from traditional teachings. Patients will be told that the study compares two training programs. To the extent possible, outcome assessors will be blinded to study arm when performing follow-up. The statistician performing the primary outcome analyses will be blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care training (Active Comparator): A refresher training course will be the equivalent of 'enhanced' usual care. Enhanced because the course will likely augment short-term knowledge of smoking cessation treatments, and participation in the study could trigger more discussions about smoking cessation than routine practice. However, it will be impossible to have any blinding between groups without at least some training.
  Interventions: Behavioral: Refresher course
- Intervention training (Experimental): The training course and decision aid aim to make treatment of tobacco use the default choice
  Interventions: Behavioral: Training program and decision aid

INTERVENTIONS:
Behavioral: Training program and decision aid — 1) a one-time, in-person, 2.5-hour training program encouraging participating GPs to present quitting smoking with a quit aid as the default choice to their eligible patients, and 2) access to an electronic decision aid that presents available quit aids. The 2.5-hour training program consists of: 1.5 hours of didactic teaching, with information about pharmacologic quit aids, electronic cigarettes, presenting quitting as a default choice, the decision aid, and a video of a model consultation. This is followed by 1 hour of role plays to practice presenting quitting as a default choice using the decision aid.
  Arms: Intervention training
Behavioral: Refresher course — A 45-minute refresher training about smoking cessation that does not aim to change GP behaviour. It will include the same information about pharmacologic quit aids and electronic cigarettes.
  Arms: Usual care training

SUMMARY:
The FIRST cluster randomized trial will evaluate the effect of 1) a training program encouraging general practitioners to offer smoking cessation treatment as a default choice to all current smokers consulting a general practitioner (GP), and 2) an interactive, electronic decision aid to guide smoking cessation treatment, on the proportion of current smokers seen in primary care who have quit smoking 6 months after a baseline visit to their GP, as compared to enhanced usual care.

DETAILED DESCRIPTION:
Smoking cessation medications are underused in primary care, likely because general practitioners (GP) lack detailed knowledge about prescribing and the fact that smokers seen in primary care must "opt-in" to treatment. Currently GPs only offer treatment to patients who say they are ready to quit smoking and desire treatment, making the default choice no treatment. Those who are not ready to quit or are hesitant do not discuss quitting or learn about options to help them quit. Further, GPs often lack confidence to discuss smoking cessation medications or do not provide patients with a choice. A decision aid can both help to present quitting with a medication as the default choice and promote shared decision making by allowing patients to see the menu of options available.

The current study will combine the use of 'default choices' when approaching smokers and shared decision making with a decision aid for choosing between smoking cessation treatments. The investigators will train GPs to offer smoking cessation as the default choice while involving patients in key decisions using a decision aid. This innovative approach has not been tested in primary care and has the potential to increase the number of current smokers who make a quit attempt with a proven quit aid, thereby increasing the number of patients who quit smoking.

The investigators will implement the training as part of the Vivre sans tabac programme for GPs run by the Swiss Medical Association (FMH).

ELIGIBILITY:
Patient-level inclusion criteria:

* Consider the GP they are seeing in consultation to be their primary care doctor
* Use tobacco daily (cigarettes, cigars, smokeless tobacco)
* ≥18 years of age at the time of inclusion

Patient-level exclusion criteria:

* Consulting for an urgent complaint that precludes even a brief discussion of smoking cessation
* Inability to follow the procedures of the study, e.g. unable to read French-language consent materials, severe psychiatric disorders, dementia, etc.
* Previous enrolment in a smoking cessation trial <1 year prior
* Current daily user of a pharmacologic smoking cessation aid

GP-level inclusion criteria:

* GP in private practice in French-speaking Switzerland (Vaud, Geneva, Jura, Neuchâtel, Fribourg or Valais) or metropolitan France
* Primarily French-speaking patients with >80 individual patients seen in a typical month

GP-level exclusion criteria:

* Completed an intensive smoking cessation curriculum <2 years prior (ie. at least half-day of training)
* Have plans to retire or relocate outside of Switzerland or France in <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 6 months follow-up after the baseline visit with a General Practitioner
  Self-reported, 7-day point-prevalence smoking abstinence

SECONDARY OUTCOMES:
Exhaled Carbon monoxide - patient | 6 month follow-up
  Chemical confirmation of abstinence among those who report 7-day smoking abstinence
Continuous abstinence - patient | 6 month follow-up
  Self-reported continuous abstinence from the patient's quit date among those who report 7-day smoking abstinence
Smoking cessation - patient | 3 weeks and 3 months follow-up
  Self-reported, 7-day point-prevalence smoking abstinence
Quit attempts - patient | 6 month follow-up
  Self-reported quit attempts (periods of abstinence to try to quit smoking) since the baseline visit
Use of quit aids - patient | 6 month follow-up
  Self-reported use of a quit aid (pharmacologic, electronic cigarette, or additional medical visits to discuss quitting) since the baseline visit
Patient participation - patient | 3 weeks follow-up
  Patient-reported participation in discussions about smoking cessation as measured by the CollaboRATE scale

OTHER OUTCOMES:
Prescribing quit aids - general practitioner | After the training program (intention), at the end of patient recruitment, and at 12-months follow-up
  The proportion of current smokers who are proposed a smoking cessation aid, as reported by GPs
Default choice approach - general practitioner | After the training program (intention), at the end of patient recruitment, and at 12-months follow-up
  Self-reported use of the default choice approach for smoking cessation
Use of decision aid - general practitioner | After the training program (intention), at the end of patient recruitment, and at 12-months follow-up
  Self-reported use of the decision aid (electronic or paper)
Discontinuation rate - GP implementation outcome | 12 months after training
  Number of GPs who recruit at least 20 patients / number of GPs randomized
Recruitment rate - patient implementation outcome | 12 months after training
  Number of patients who sign consent / number of patients provided information about the trial
Discontinuation rate - patient implementation outcome | 12 months after training
  Number of patients who complete 6-month follow-up / number of patients who sign consent

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Selby, MD, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Locations (2):
- Maison de santé Mermoz, Lyon, France
- Unisante, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Anonymised data available upon request

REFERENCES:
- [Background] Jakob J, Cornuz J, Auer R, Jacot Sadowski I, Cardinaux R, Selby K. [Design and user-testing of a decision aid comparing medications for smoking cessation]. Rev Med Suisse. 2017 Jun 7;13(566):1191-1194. French. PMID 28640564
- [Background] Hempel-Bruder C, Habfast-Robertson I, Durand MA, Berlin I, Marti J, Khazaal Y, Quinto C, Faouzi M, Selby K. Combining default choices and an encounter decision aid to improve tobacco cessation in primary care patients: protocol for a cluster-randomized trial. BMC Prim Care. 2022 Sep 24;23(1):246. doi: 10.1186/s12875-022-01859-9. PMID 36151529
- [Derived] Selby K, Habfast-Robertson I, Durand MA, Hempel-Bruder C, Boesch A, Marti J, Kazaal Y, Faouzi M, Maisonneuve H, Berlin I. Combining Default Choices and an Encounter Decision Aid to Improve Tobacco Cessation in Primary Care Patients: A Pragmatic, Cluster-Randomized Trial. J Gen Intern Med. 2025 Sep;40(13):3078-3085. doi: 10.1007/s11606-024-09088-9. Epub 2024 Oct 9. PMID 39384691
- See also: Electronic decision aid used in trial — http://howtoquit.ch
- See also: Paper decision aid used in trial — https://www.unisante.ch/sites/default/files/inline-files/UNI_tableau_stop_tabac-compressed.pdf